CLINICAL TRIAL: NCT01358344
Title: A Study to Determine the Bioequivalence of SCH 530348 2.5 mg Tablets Containing a High and Low Percentage of Drug as the Free Base Within the Range Used in the Pivotal Phase 3 Efficacy and Safety Trials. (Protocol No. P06558)
Brief Title: A Bioequivalence Study of SCH 530348 2.5 mg Tablets (P06558)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P06558
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Pantoprazole; vorapaxar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Percentage (Experimental)
  Interventions: Drug: Pantoprazole; Drug: SCH 530348 (standard percentage)
- High Percentage (Experimental)
  Interventions: Drug: Pantoprazole; Drug: SCH 530348 (high percentage)

INTERVENTIONS:
Drug: Pantoprazole — 40 mg delayed-release tablet administered orally in the morning of Days 1-7
Drug: SCH 530348 (high percentage) — 2.5 mg tablet containing ~46% active pharmaceutical ingredient (API) as free base (46+5%) administered orally on the morning of Day 5
  Arms: High Percentage
Drug: SCH 530348 (standard percentage) — 2.5 mg tablet containing ~23% API as free base (STANDARD) administered orally on the morning of Day 5
  Arms: Standard Percentage

SUMMARY:
The purpose of this study is determine if SCH 530348 2.5 mg tablets containing a high percentage of drug as the free base are equivalent to tablets with the standard percentage when given to participants.

ELIGIBILITY:
Inclusion criteria:

* Body Mass Index (BMI) between 18 and 32, inclusive
* Clinical laboratory tests within normal limits
* Free of any clinically significant disease that would interfere with the study evaluations
* Screening 12-lead electrocardiogram (ECG) conduction intervals within gender-specific normal range
* Vital sign measurements within the following ranges: oral body temperature, 35.0°C to 37.5°C; systolic blood pressure, 90 to 140 mmHg; diastolic blood pressure, 45 to 90 mmHg; pulse rate, 40 to 100 beats per minute
* Female participants must be postmenopausal, surgically sterile, abstinent, or using medically accepted method of contraception for 3 months prior to the screening period, during the trial, and for 2 months after stopping the trial. Non-vasectomized men must agree to use acceptable contraception or to abstain from sexual intercourse during the trial and for 3 months after stopping the medication

Exclusion Criteria:

* Female participants who are pregnant, intend to become pregnant (within 3 months of ending the study), or are breastfeeding
* History of coagulation disorder(s), thrombocytopenia, bleeding tendency, ulcers, or gastrointestinal bleeding
* History of cardiac abnormalities including clinically relevant ECGs, frequent palpitations or syncopal episodes
* Any surgical or medical condition that might significantly alter the absorption, distribution, metabolism or excretion of any drug
* History of any infectious disease within 4 weeks prior to drug administration
* Positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV)
* Positive screen for drugs with a high potential for abuse
* History of alcohol or drug abuse in the past 2 years
* Blood donation in the past 60 days
* Previous treatment with SCH 530348
* Currently participating in another clinical study or has participated in a clinical study within 30 days
* Demonstrated allergic reactions
* Smokes more than 10 cigarettes or equivalent tobacco use per day
* History of malignancy
* Has received any protocol-defined treatment which could interfere with ability to participate in the trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from 0 to 72 hours (AUC[0-72h]) of SCH 530348 | Up to 72 hours after SCH 530348 dose on Day 5
Maximal plasma concentration (Cmax) of SCH 530348 | Up to 72 hours after SCH 530348 dose on Day 5

SECONDARY OUTCOMES:
Number of participants experiencing clinical and laboratory adverse events (AEs) | Up to 2 weeks after last dose